CLINICAL TRIAL: NCT00979940
Title: Effects of Short Term, High Dose Atorvastatin Therapy on Periprocedural Myonecrosis and Platelet Inhibition After PCI
Brief Title: Effects of Short Term, High Dose Atorvastatin Therapy on Periprocedural Myonecrosis and Platelet Inhibition After Percutaneous Coronary Intervention (PCI)
Acronym: ESTATE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slower than anticipated enrollment for pilot study.
Sponsor: Indiana University School of Medicine (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0712-15; 1470
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2015-09-22 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-08

CONDITIONS: Coronary Artery Disease
Keywords: atorvastatin; clopidogrel; percutaneous intervention; periprocedural myonecrosis
MeSH Terms: conditions — Coronary Artery Disease | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No atorvastatin (No Intervention): Patients do not receive Atorvastatin prior to PCI in cath lab
- atorvastatin (Experimental): Atorvastatin 80mg po given prior to PCI in cath lab
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 80mg po given one time before PCI in cath lab.
  Arms: atorvastatin

SUMMARY:
This research study plans to evaluate the use of atorvastatin in patients with coronary artery disease given immediately before PCI and whether it will decrease the amount of heart damage after PCI.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing revascularization for significant coronary artery disease
* age range 21-85 years

Exclusion Criteria:

* non-STEMI, STEMI
* cancer
* renal failure with creatinine>3.0mg/dl
* liver cirrhosis
* lymphoproliferative disorder
* pregnancy
* thrombocytopenia<150'000
* coagulopathy (INR>1.5)
* abnormal liver function tests
* illicit drug use
* history of statin intolerance
* history of rhabdomyolysis
* planned use of Glycoprotein IIb/IIIa inhibitors during PCI
* current therapy with atorvastatin, pravastatin, lovastatin, fluvastatin, or rosuvastatin

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-11; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Kreutz, MD, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Methodist Hospital, Indianapolis, Indiana
  - Wishard Hospital, Indianapolis, Indiana

REFERENCES:
- [Derived] Kreutz RP, Breall JA, Sinha A, von der Lohe E, Kovacs RJ, Flockhart DA. Simultaneous administration of high-dose atorvastatin and clopidogrel does not interfere with platelet inhibition during percutaneous coronary intervention. Clin Pharmacol. 2016 Jun 3;8:45-50. doi: 10.2147/CPAA.S98790. eCollection 2016. PMID 27350760

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Atorvastatin | Atorvastatin
Started | 32 | 28
Completed | 32 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Atorvastatin | Atorvastatin | Total
Number analyzed (Participants) | 32 | 28 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (8) | 62.6 (10) | 61.9 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 25 | 22 | 47

OUTCOME MEASURES:

1. Primary Outcome: Periprocedural Myonecrosis
Time Frame: 16-24 hours post PCI
Measure: Number; unit: participants
Arm/Group | No Atorvastatin | Atorvastatin
Number analyzed (Participants) | 32 | 28
participants | 17 | 15
Statistical Analysis 1: Comparison: No Atorvastatin vs Atorvastatin; Test type: Superiority or Other; p = 0.97, Chi-squared

ADVERSE EVENTS:
Arm/Group | No Atorvastatin | Atorvastatin
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/28
Other Adverse Events (participants affected / at risk) | 0/32 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No